CLINICAL TRIAL: NCT02137083
Title: A Prospective Single-center Randomized Phase 2 Trial Comparing Docetaxel Plus Fulvestrant With Docetaxel in Postmenopausal, Hormone-receptor Positive and HER2-negative Metastatic Breast Cancer
Brief Title: A Trial Comparing Docetaxel Plus Fulvestrant With Docetaxel in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Vice Director of department of medical oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2014-13
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Chemotherapy; Endocrine therapy; Docetaxel; Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel Plus Fulvestrant (Experimental): Docetaxel:75mg/m2 D2 every 21 days
  Fulvestrant:500mg D1, D15, D29, D57, every 28 days later
  Interventions: Drug: Docetaxel; Drug: Fulvestrant
- Docetaxel (Active Comparator): Docetaxel:75mg/m2 D2 every 21 days
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — 75mg/m2 D2 every 21 days
  Other Names: Taxotere
Drug: Fulvestrant — 500mg D1, D15, D29, D57, every 28 days later
  Other Names: Faslodex
  Arms: Docetaxel Plus Fulvestrant

SUMMARY:
Comparing Docetaxel Plus Fulvestrant With Docetaxel in Patients With Metastatic Breast Cancer

DETAILED DESCRIPTION:
Comparing Docetaxel Plus Fulvestrant With Docetaxel in Postmenopausal, Hormone-receptor Positive and HER2-negative Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female between 18 and 70 years old
* ECOG performance status of ≤ 1
* Life expectancy more than 3 months
* Histologically confirmed metastatic breast cancer
* ER and&or PR pqositive, HER2-negative
* Disease progression during adjuvant or first-line endocrine therapy, or endocrine naive but unsuitable for endocrine therapy alone
* No pretreated chemotherapy for metastatic disease
* Have at least one target lesion according to RECIST 1.1
* No therapy (chemotherapy, endocrine therapy, target therapy and operation) within 4 weeks before enrollment
* Hemoglobin ≥ 90 g/L, Absolute Neutrophil Count ≥ 1.5×10^9/L, Platelet Count ≥ 75×10^9/L, Serum Bilirubin ≤ 1.5×ULN, ALT and AST ≤ 1.5×ULN, Serum Creatinine ≤ 1×ULN, Endogenous Creatinine Clearance>50ml/min

Exclusion Criteria:

* Pregnant or lactating women
* Evidence of CNS metastasis
* Seriously uncontrolled infection
* History of another malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pretreated with Fulvestrant
* Pretreated with two or more lines of endocrine therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 6 weeks

SECONDARY OUTCOMES:
Overall Response Rate | 6 Weeks
Overall Survival | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China